CLINICAL TRIAL: NCT01400191
Title: The Inhibitory Effect of Metformin on Gluconeogenesis in Relation to Polymorphisms in Organic Cation Transporter 1 (OCT1) in Healthy Volunteers
Brief Title: The Inhibitory Effect of Metformin on Gluconeogenesis in Relation to Polymorphisms in Organic Cation Transporter 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Mette Marie Hougaard Christensen, MD, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AKF 379
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Pharmacogenetics of Metformin
Keywords: Metformin; Hypoglycemic Agents; Diabetes Mellitus, Type 2; Gluconeogenesis; Pharmacodynamics; Pharmacogenetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Homozygote wildtype OCT1 (Active Comparator)
  Interventions: Drug: Metformin
- Heterozygote OCT1 (Active Comparator)
  Interventions: Drug: Metformin
- Homozygote OCT1 variant (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — The study was designed as a randomized, cross-over trial with a washout period of at least 4 weeks between the phases. In both phases, the volunteers fasted for 42 h. This was done in order to include an evaluation of the pharmacodynamic effect of metformin on the glucose production in fasting healthy volunteers.

SUMMARY:
The aim of the study is to evaluate the pharmacodynamic impact of metformin in healthy Caucasian volunteers with and without single polymorphisms M420del or R61C in OCT1, thus the study hypothesis is that metformin only affect the hepatic gluconeogenesis in healthy volunteers with functional OCT1-transporters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Written consent
* Genotyped in OCT1 for (M420del and R61C)

Exclusion Criteria:

* Daily medication
* Alcohol abuse
* Pregnancy
* Breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Endogenous glucose production | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mette Marie H Christensen, MD, Principal Investigator — Department of Public Health, Clinical Pharmacology, University of Southen Denmark
Locations (1):
- Clinical pharmacology, Institute og public health, University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Derived] Christensen MM, Hojlund K, Hother-Nielsen O, Stage TB, Damkier P, Beck-Nielsen H, Brosen K. Endogenous glucose production increases in response to metformin treatment in the glycogen-depleted state in humans: a randomised trial. Diabetologia. 2015 Nov;58(11):2494-502. doi: 10.1007/s00125-015-3733-2. Epub 2015 Aug 14. PMID 26271344